CLINICAL TRIAL: NCT05366660
Title: Remote Programming of Cardiac Implantable Electronic Device
Acronym: REACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2021/07
Record Dates: First submitted 2022-05-05; First posted 2022-05-09 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Defibrillators, Implantable; Follow-Up Studies; Pacemaker, Artificial; Telemedicine; Algorithms
Keywords: Implantable cardioverter defibrillator; ICD; Pacemaker; Telemedicine; Remote monitoring; Cardiac implantable electronical device

STUDY DESIGN:
Intervention Model Description: Multicenter feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CIED's interrogation/programming (Experimental): All the patients will be included in this single arm to interrogate/programm their CIED
  Interventions: Other: Interrogation/programming

INTERVENTIONS:
Other: Interrogation/programming — As the study investigates remote programming, we will describe two locations: local (patient side) and remote (expert side). Local support is defined by a physician or a technician under the direct responsibility of a nearby physician who connect the patient to the remote programming system. Similar to a conventional check-up, an external defibrillator will be located in the near vicinity of the patient. The patient will first be connected to the programmer as during a conventional follow-up. The programmer will then be connected to a local PC which captures the programmer VGA video output and controls the programmer through a mouse emulator. This local PC will be remotely controlled by the remote PC using Cisco Webex, a communication software used worldwide to support telemedicine.

SUMMARY:
Cardiac Implantable Electronic Devices (CIEDs) such as pacemakers and implantable cardioverter defibrillators, need to be regularly interrogated and reprogrammed to ensure proper functioning. While remote monitoring allows for partial interrogation at a remote location, full interrogation and changing the CIED parameters is only possible when the patient visits a cardiologist capable of performing device programming. This can be challenging for patients and may cause unnecessary delays, particularly in settings of limited resources, enforced physical distancing, and quarantines. We aim to investigate the efficacy and safety of remote programming.

DETAILED DESCRIPTION:
Cardiac Implantable Electronic Devices (CIEDs) such as pacemakers and implantable cardioverter defibrillators, need to be regularly interrogated to guarantee proper functioning. In France, the follow-up of approximately 400 000 patients implanted with a CIED is performed by cardiologists. Remote monitoring allows for interrogation of contemporary CIEDs and has revolutionized the care for implanted patients. Early detection of arrhythmias, lead issues, battery depletion and algorithm side effects decreases both morbidity and mortality of CIED patients which is why today remote monitoring enjoys a class IA recommendation. While remote interrogation is advancing steadily, remote programming is not at all possible today. CIED problems may be quickly solved by changing the parameters but this is only possible when the patient visits a cardiologist capable of performing CIED programming. This can be challenging for patients and may cause unnecessary delays, particularly in settings of limited resources, enforced physical distancing, and quarantines. Remote programming of a CIED offers multiple advantages such as shorter travel distances for the patient, reduced need for presence of specialized cardiologists (in small clinics or diagnostic centers) and the possibility to offer expert support at remote locations or developing countries. At Bordeaux University, we have developed a method which enables remote programming of a CIED. The method requires the patient to be in direct vicinity of a CIED programmer, while the cardiologist specialized in CIED programming can operate the programmer from any remote location. We aim to investigate the efficacy and safety of remote programming by applying our method to implanted patients to perform remote interrogation and programming changes.

ELIGIBILITY:
Inclusion Criteria:

* Patient of both sexes over the age of 18
* Patients implanted with a cardiac pacemaker or an automatic defibrillator and an indication for device check-up (interrogation ± programming) which may be periodic as part of their follow-up, postoperative, following a remote monitoring alert, pre/post MRI or following symptoms.
* Person beneficiary of social security insurance.
* Informed consent confirmed in writing (at the latest on the day of inclusion and before any examination required by the research).
* Women of procreating age with effective contraception

Exclusion Criteria:

* Patients younger than 18 years old
* Patients who are incapable to understand the study design or to give informed consent.
* Pregnant or breastfeeding women
* Persons placed under judicial protection, curatorship, tutorship.
* Subject deprived of liberty on judicial or administrative decision
* Persons participating in another study who are still in their period of exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Successful remote interrogation and programming of CIED | 18 months
  Success rate of remote interrogation and programming of CIED

SECONDARY OUTCOMES:
To assess the user-friendliness of the system (1) | 18 months
  Time of the procedure (interrogation and programming)
To assess the user-friendliness of the system (2) | 18 months
  Type of programming modifications done
To assess the user-friendliness of the system (3) | 18 months
  Time of intallation procedure
To assess the user-friendliness of the system (4) | 18 months
  Turnaround time of the command

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain MD Ploux, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Bordeaux University Hospital, Pessac, France, France